CLINICAL TRIAL: NCT06511440
Title: Assessment of an Automated Optical Coherence Tomography and Camera : Reference Database
Status: Completed | Type: Observational
Sponsor: Crystalvue Medical Coporation (Industry)
Responsible Party: Sponsor
Other Study IDs: Vision-700 Reference database
Record Dates: First submitted 2024-07-04; First posted 2024-07-22 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy group: Subject without eye disease
  Interventions: Device: Vision-700

INTERVENTIONS:
Device: Vision-700 — OCT machines used for diagnostic purposes

SUMMARY:
The objective of this study is to establish the Reference database of Vision-700.

DETAILED DESCRIPTION:
The objective is to collect and establish the Reference database of Vision-700, which is expected to recruit subjects with normal vision to collect the optical coherent tomography measurement data.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects 22 years of age or older on the date of informed consent
2. Subjects able to understand the written informed consent and willing to participate as evidenced by signing the informed consent
3. Subjects presenting at the site with normal eyes bilaterally
4. IOP ≤ 21 mmHg bilaterally
5. BCVA 20/40 or better bilaterally

Exclusion Criteria:

1. Subjects unable to tolerate ophthalmic imaging.
2. Subjects with ocular media not sufficiently clear to obtain acceptable OCT images.
3. HFA visual field (24-2 Sita Standard, white on white) result unreliable (based on manufacturer's recommendation), defined as fixation losses > 20% or false positives > 33%, or false negatives > 33%
4. Visual field defects consistent with glaucomatous optic nerve damage based on at least one of the following two findings: On pattern deviation (PD), there exists a cluster of 3 or more points in an expected location of the visual field depressed below the 5% level, at least 1 of which is depressed below the 1% level; Glaucoma hemi-field test "outside normal limits."
5. History of leukemia, dementia or multiple sclerosis.
6. History of hydroxychloroquine or chloroquine use.
7. Subjects with photosensitivity.
8. Subject having Photodynamic therapy (PDT) within 6 months.
9. Subjects taking photosensitivity drug currently.

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy subjects
Sampling Method: Non-Probability Sample
Enrollment: 285 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
The reference OCT data | 2022/09/01
  The study is to collect OCT measurement data on normal healthy eyes in order to establish the reference data range for OCT parameters, included full retinal thickness (μm), retinal nerve fiber layer (μm), ganglion cell complex thickness (μm) and optic nerve head (μm). The reference data range will provide it with the doctor to dignoisis.

CONTACTS AND LOCATIONS:
Overall Officials: Liang I-Chia, Principal Investigator — Tri-Services General Hospital
Locations (1):
- Tri-Services General Hospital, Taipei County, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided